CLINICAL TRIAL: NCT05030467
Title: Leveraging Electronic Health Record (EHR) Tools to Reduce Health Disparities for Patients With Uncontrolled Hypertension
Acronym: REDUCE-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002479; R01MD014874 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Providers within the clinics randomized to the intervention arm will receive a variety of EHR-based tools for eligible patients with uncontrolled hypertension.
  Interventions: Behavioral: REDUCE-BP Intervention
- Control Arm (No Intervention): Providers within the clinics randomized to usual care will receive no EHR tools, except those currently available in clinical practice.

INTERVENTIONS:
Behavioral: REDUCE-BP Intervention — Pre-visit:
  Providers in the intervention arm will receive dashboards which will highlight racial/ethnic differences in rates of achieving blood pressure control within their patient panel. The dashboard will also provide individual-level information for patients with poorly controlled blood pressure.
  During visit:
  Providers will receive clinical decision support within relevant patients' charts that highlight the patient's under-treated blood pressure and potential impacts of social needs.
  Providers will have the opportunity to provide enhanced patient education materials, which can be automatically ordered within the clinical decision support.
  Post-visit:
  Patient-subjects' access to the online patient portal will be streamlined by the inclusion of information about the patient portal in the patients' after-visit summary. Providers will also be able to referral patients automatically to nurse BP visits.
  Arms: Intervention Arm

SUMMARY:
A two-arm cluster randomized controlled trial targeting primary care providers will be conducted to evaluate the impact of a multicomponent electronic health record (EHR) intervention on hypertension management. Given the cluster trial design, randomization will be conducted at the site level, and in the intervention sites, all eligible providers will receive the intervention. The intervention consists of enhancing tools already available to primary care providers in the EHR system, including developing and implementing provider disparities dashboards, enhancing electronic decision support, and simplifying self-monitoring orders and communication materials. The intervention aims to improve blood pressure control and reduce health disparities in racial and ethnic minorities. Findings from this trial will provide important insight into whether a multicomponent intervention targeting providers and leveraging health information technology can reduce health disparities.

DETAILED DESCRIPTION:
The goal of this project is to improve existing decision support for hypertension control and to reduce disparities in treatment, consistent with Advocate-specific professional guidelines and quality metrics. To achieve this, a cluster randomized trial will be conducted and evaluated to determine whether health IT tools targeted to providers improve blood pressure control for patients with uncontrolled hypertension.

The primary hypothesis is that a health IT intervention will improve systolic blood pressure (primary outcome), concordance with hypertension guidelines (secondary outcome), diastolic blood pressure (secondary outcome), treatment intensification (secondary outcome), controlled blood pressure (secondary outcome) and systolic blood pressure disparities (secondary outcome) compared with usual care.

Participating clinics will be randomly assigned to one of 2 arms: (a) Arm 1: multicomponent, intervention and (b) Arm 2: usual care (i.e. no intervention). Providers and in each arm will receive the same intervention for up to 24 months after randomization, which will demonstrate the relative effectiveness of each approach as well as its long-term impact on clinical outcomes. Primary care providers in the intervention clinics will receive electronic decision support tools to guide their care of eligible patients. Providers in usual care clinics will receive usual care at Advocate Aurora Health (AAH). Patients will not receive any intervention or outreach independent of their provider or care team. EHR data will be used to implement the EHR tools, identify study subjects, track study progress, and evaluate the effect of the interventions. Patients will only be included in the analysis and will not be directly enrolled or contacted by investigators; we expect at least 2000 patients to be included in the analysis.

ELIGIBILITY:
24 practices will be randomized to either Intervention or Control. We will include in the analysis patients who meet the following Inclusion Criteria:

1. Medical Group Medical Home Population: 1 visit with Primary Care Physician (PCP) in past 2 years (rolling 24 months) and Patient has a medical group PCP as their EPIC General PCP
2. Current age 18-85 years
3. Hypertension diagnosis on EPIC Problem list OR at least 2 visits (office/telehealth/telephonic) with an encounter diagnosis of hypertension on different dates, with any during the last 24 months (rolling dates) performing provider
4. Latest outpatient/ambulatory (exclude urgent care) systolic blood pressure ≥140 or diastolic blood pressure ≥90 (12 months rolling) (lowest measure if more than one taken at the same time)

Exclusion Criteria:

* Patients not meeting the inclusion criteria above will not be included in the analysis of the study. No other exclusion criteria will be used.

Among these eligible patients, patients included in the primary analysis will be those that had an in-person visit at one of the trial clinics.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49210 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Advocate Health Care, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 clinics were randomized to intervention and control (1:1). Patients were identified from EHR data on the basis of their meeting eligibility criteria at the randomized clinics. Providers from these clinics were not directly enrolled in the study. Outcomes were measured at the patient level.
Units Other Than Participants: Clinics
Groups:
- Intervention Arm: Providers within the clinics randomized to the intervention arm will receive a variety of EHR-based tools for eligible patients with uncontrolled hypertension.
  REDUCE-BP Intervention: Pre-visit:
  Providers in the intervention arm will receive dashboards which will highlight racial/ethnic differences in rates of achieving blood pressure control within their patient panel. The dashboard will also provide individual-level information for patients with poorly controlled blood pressure.
  During visit:
  Providers will receive clinical decision support within relevant patients' charts that highlight the patient's under-treated blood pressure and potential impacts of social needs.
  Providers will have the opportunity to provide enhanced patient education materials, which can be automatically ordered within the clinical decision support.
  Post-visit:
  Patient-subjects' access to the online patient portal will be streamlined by the inclusion of information about the patient portal in the patients' after-visit summary. Providers will also be able to referral patients automatically to nurse BP visits.
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 24747; 12 Clinics | 24463; 12 Clinics
Completed | 24747; 12 Clinics | 24463; 12 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: This is the number of patients who met eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 24747 | 24463 | 49210
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (12.5) | 64.7 (12.5) | 64.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14977 | 14143 | 29120
  Male | 9770 | 10320 | 20090
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2922 | 1929 | 4851
  Not Hispanic or Latino | 21079 | 21890 | 42969
  Unknown or Not Reported | 746 | 644 | 1390
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 162 | 213 | 375
  Asian | 1093 | 1458 | 2551
  Native Hawaiian or Other Pacific Islander | 173 | 127 | 300
  Black or African American | 13997 | 10803 | 24800
  White | 8291 | 11137 | 19428
  More than one race | 126 | 127 | 253
  Unknown or Not Reported | 905 | 598 | 1503
Baseline systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 145.4 (14.3) | 145.3 (14.3) | 145.4 (14.3)
Baseline diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 80.4 (10.8) | 80.6 (10.7) | 80.5 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from identification to the end of the 12-month follow-up, using values in the EHR from ambulatory care encounters
Time Frame: 12 months
Population: Patients identified as eligible were included in the analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 24747 | 24463
mmHg | -11.0 (19.2) | -11.0 (19.1)
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; We used generalized estimating equations (GEE) to adjust for the cluster design with an identify link function and normally-distributed errors; Test type: Superiority; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.39 to 0.31]

2. Secondary Outcome: Percentage of Patients With Well-controlled Blood Pressure
Description: Percentage of patients with well-controlled blood pressure (<140/90mmHg) in the 12-month follow-up period, using values in the EHR from ambulatory care encounters
Time Frame: 12 months
Population: Patients identified as eligible were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 24747 | 24463
Participants | 16910 | 16441
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Outcomes were evaluated using generalized estimating equations with a log link and Poisson-distributed errors, adjusting for clinic-level clustering; Test type: Superiority; p = 0.011, Regression, Logistic; Risk Ratio (RR) = 1.02, 95% CI 2-sided [1.00 to 1.03]

3. Secondary Outcome: Percentage of Patients With Intensification of Medication
Description: Percentage of patients with intensification of medication in the 12-month follow-up period, defined by addition of therapy or increasing dose.
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Patients With Guideline-concordant Medications
Description: Percentage of patients with guideline-concordant medications ordered in the follow-up period
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from identification to 12-month follow-up, measured using values in the EHR
Time Frame: 12 months
Population: Patient identified as eligible for analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 24747 | 24463
mmHg | -4.4 (10.8) | -4.3 (10.9)
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.383, Regression, Linear; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.38 to 0.15]

6. Secondary Outcome: Systolic Blood Pressure Differences
Description: Change in the gap in systolic blood pressure (SBP) between Black and White patients and Hispanic/Latino and Non-Hispanic/Latino patients from identification to the end of the 12-month follow-up, measured using values in the EHR from ambulatory care encounters
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Description: Deaths and adverse events are reported for intervention clinic patients who were included in the analyses for the trial; information was not collected on control clinic patients. We used an automatic adverse event reporting system to monitor for any AEs that occurred, which were routinely reviewed by quality and safety specialists at the institution. For deaths, we identified patient deaths through a retrospective review within the EHR based on reports.
Groups:
- Control Arm - Not Collected for the Adverse Event Reporting: Providers within the clinics randomized to usual care will receive no EHR tools, except those currently available in clinical practice.
  Information on control clinic patients was not collected as part of the adverse event reporting.
Arm/Group | Intervention Arm | Control Arm - Not Collected for the Adverse Event Reporting
All-Cause Mortality (participants affected / at risk) | 3/24747 | 0/0
Serious Adverse Events (participants affected / at risk) | 24/24747 | 0/0
Other Adverse Events (participants affected / at risk) | 17/24747 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=24747) | Control Arm - Not Collected for the Adverse Event Reporting (N=0)
Unrelated SAE (Blood and lymphatic system disorders) | 24 (24) | 0 (0) — All SAEs were deemed unrelated to the intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=24747) | Control Arm - Not Collected for the Adverse Event Reporting (N=0)
Unrelated AE (Blood and lymphatic system disorders) | 17 (17) | 0 (0) — All AEs were deemed unrelated to the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05030467/Prot_SAP_000.pdf